CLINICAL TRIAL: NCT00987818
Title: Reduction of Antibiotic Use in the ICU: Procalcitonin Guided Versus Conventional Antibiotic Therapy in Patients With Sepsis in the ICU
Brief Title: Procalcitonin Guided Versus Conventional Antibiotic Therapy in Patients With Sepsis in the ICU
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No MEC approval
Sponsor: Rijnstate Hospital (Other)
Collaborators: Stichting Vrienden van het Alysis Leerhuis (Unknown)
Responsible Party: HJ van Leeuwen, MD PhD, Alysis Zorggroep, Rijnstate Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 630-190809
Record Dates: First submitted 2009-09-16; First posted 2009-10-01 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2012-12

CONDITIONS: Sepsis; Intensive Care
Keywords: Biomarkers; Antibiotic therapy
MeSH Terms: conditions — Sepsis | interventions — Procalcitonin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- PCT guided antibiotic therapy (Experimental)
  Interventions: Other: Procalcitonin measurement
- Standard antibiotic therapy (Placebo Comparator)
  Interventions: Other: Procalcitonin measurement

INTERVENTIONS:
Other: Procalcitonin measurement — Daily procalcitonin measurement. Antibiotic discontinuation policy dependent on procalcitonin value. In the control group standard duration of antibiotic therapy.

SUMMARY:
The adequacy of early empiric antimicrobial therapy is an important factor in determining the outcome in patients with severe sepsis. The duration of adequate antibiotic therapy in these patients however is less clear. Duration of antibiotic therapy in patients with sepsis in the ICU based on inflammatory markers has not been extensively studied.

Procalcitonin (PCT) is an acute phase protein that has prognostic value in critically ill patients and can be used to monitor disease activity in sepsis and systemic inflammation. This study will examine the effect of PCT guided antibiotic therapy compared with conventional antibiotic therapy on treatment duration in patients with sepsis admitted to the ICU.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the ICU
* Age > 18 years
* Antibiotic therapy for sepsis with a suspected or proven focus of infection

Exclusion Criteria:

* Age < 18 years
* Pregnancy
* Infection or presumed infection requiring prolonged antibiotic therapy (osteomyelitis, meningitis, endocarditis, septic arthritis, mediastinitis, tuberculosis, Pneumocystis jiroveci pneumonia, Toxoplasmosis, Legionellosis, Listeriosis)
* Indication for prolonged systemic prophylactic antibiotic therapy
* Severe viral or parasitic infections (hemorrhagic fever, malaria)
* Antibiotic therapy started 48 hours before enrollment
* Severe immunocompromised patients (AIDS with a CD4 count < 200cells/mm3, severe neutropenia(<500 neutrophils/mm3), patients undergoing immunosuppressive therapy after solid organ transplantation)
* Patients foregoing life sustaining treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
duration of antibiotic therapy | 28 days

SECONDARY OUTCOMES:
28 day mortality | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Alysis Zorggroep, Rijnstate Hospital, Arnhem, Gelderland, Netherlands